CLINICAL TRIAL: NCT00388479
Title: A Multicenter Phase III, Double-Blind, Placebo-Controlled, Parallel Study of ADL-8-2698 in Opioid-Induced Postoperative Bowel Dysfunction/Postoperative Ileus
Brief Title: Study of Alvimopan for the Management of Opioid-induced Postoperative Bowel Dysfunction/ Postoperative Ileus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14CL308
Record Dates: First submitted 2006-10-12; First posted 2006-10-16 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2015-07

CONDITIONS: Ileus
MeSH Terms: conditions — Ileus | interventions — alvimopan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Alvimopan

SUMMARY:
Patients undergoing major abdominal surgery are at highest risk for developing postoperative ileus (POI), occurring in nearly all cases. Signs and symptoms of POI may include abdominal distention and bloating, persistent abdominal pain; nausea and/or vomiting; delayed passage or inability to pass flatus or stool; and inability to tolerate a solid diet. This study will test the ability of alvimopan 6 mg or 12 mg given 2 hours before the scheduled start of surgery to hasten the recovery of GI function in patients undergoing major abdominal surgery (bowel resection or abdominal hysterectomy).

DETAILED DESCRIPTION:
Postoperative ileus (POI) is a temporary slowing down or stopping of bowel function and a slowing down of movement of contents of the intestines. This functional impairment persists for a variable duration following surgery, usually resolving within 1 day in the small intestine, 1 to 3 days in the stomach and 3 to 5 days in the colon. When POI persists for more than 5 days, it is generally considered severe, sometimes referred to as complicated or prolonged POI, and increases the risk for related morbidity. No drug therapy has been shown to consistently shorten the duration of POI. This study is designed to demonstrate that alvimopan, a novel, peripherally acting mu opioid receptor antagonist, accelerates the recovery of GI function in patients undergoing bowel resection or hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled for a partial small/large bowel resection with primary anastomosis or total abdominal hysterectomy (simple or radical) via laparotomy
* Subject is scheduled to receive primary postoperative pain management with intravenous (i.v.) patient-controlled analgesia (PCA) opioids

Exclusion Criteria:

* Subject is scheduled for a total colectomy, colostomy, ileostomy
* Subject has complete bowel obstruction
* Subject has recently been on an acute course (1-10 days) of opioid analgesics and has not been off all opioids for at least 1 week prior to surgery Subject has been on chronic (>10 days) opioid analgesics and has not been off all opioids for at least 2 weeks prior to surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 666
Dates: Start 2001-12; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Acceleration of gastrointestinal recovery

SECONDARY OUTCOMES:
Time until ready for discharge based upon recovery of GI function
Severity of GI symptoms
Pain
Opioid Consumption
Time to tolerate liquids
Need for reinsertion of nasogastric tube
Time until discharge order is written

CONTACTS AND LOCATIONS:
Overall Officials: Adolor Corporation, Study Director — Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)
Locations (1):
- Various, Exton, Pennsylvania, United States

REFERENCES:
- [Result] Viscusi ER, Goldstein S, Witkowski T, Andonakakis A, Jan R, Gabriel K, Du W, Techner L, Wallin B. Alvimopan, a peripherally acting mu-opioid receptor antagonist, compared with placebo in postoperative ileus after major abdominal surgery: results of a randomized, double-blind, controlled study. Surg Endosc. 2006 Jan;20(1):64-70. doi: 10.1007/s00464-005-0104-y. Epub 2005 Dec 7. PMID 16333556
- [Derived] Ludwig K, Viscusi ER, Wolff BG, Delaney CP, Senagore A, Techner L. Alvimopan for the management of postoperative ileus after bowel resection: characterization of clinical benefit by pooled responder analysis. World J Surg. 2010 Sep;34(9):2185-90. doi: 10.1007/s00268-010-0635-9. PMID 20526599